CLINICAL TRIAL: NCT00903318
Title: Male:Female Birth Ratios and Phthalate Levels Along The Rural Lower Rio Grande Valley (Hidalgo County) and in Baytown, Texas
Brief Title: Male:Female Birth Ratios and Phthalate Levels
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2008-0742; 5P60MD000503 (NIH)
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Endocrine Diseases
Keywords: Endocrine; Environmental Chemicals; Male:Female Birth Ratio; Phthalate Exposure; Generational sex ratio trends; Mexican American; Baytown; Rio Grande Valley; Hidalgo County; Texas
MeSH Terms: conditions — Endocrine System Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine sample.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mexican American Men and Women: Rural and urban Mexican American men and women , aged 18 to 40, in urban Baytown, TX and rural Rio Grande Valley (Hidalgo County) communities along the Texas-Mexico border
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire about family's characteristics taking about 30-35 minutes to complete.
  Other Names: Survey

SUMMARY:
Objective 1: To assess environmental exposure to chemicals/toxins, including phthalates, among rural and urban Mexican American men and women (n=300), aged 18 to 40, in urban Baytown, TX and rural Rio Grande Valley (Hidalgo County) communities along the Texas-Mexico border region via survey.

Objective 2: To determine generational sex ratio trends in urban Baytown, TX and along the rural Rio Grande Valley (Hidalgo County) utilizing vital statistics data from the Texas Department of Health and the Center for Health Statistics.

Objective 3: To measure urinary phthalate levels and self-reported phthalate exposure in Mexican American men and women from urban Baytown, Texas and rural communities along the lower Rio Grande Valley (Hidalgo County) on theTexas-Mexico border. To conduct an optional procedure, chromosomal sex determination, among a subgroup of 50 persons (13 men + 12 women in each community) from participants who complete the survey in Objective 1.

DETAILED DESCRIPTION:
Questionnaire:

If you agree to take part in this study, you will complete a questionnaire about your family's characteristics. For example, the questionnaire will have questions about your educational level, your eating habits, your health conditions, your family's income level, and how many people live in your house. The study doctor will also ask you questions about any drugs you may be taking. The questionnaire should take about 30-35 minutes to complete.

The completed paper questionnaire will be placed in a secured, locked cabinet and will be given a code number. Only the researcher in charge of the study will have access to the code numbers and be able to link the questionnaire to you. After the study ends and after information from the questionnaire has been entered in a password protected database, the paper copy of the questionnaire will be sent to M. D. Anderson to be stored for up to 5 years. After 5 years, it will be destroyed.

Urine Sample:

You will have a urine sample collected. Researchers will study the urine samples to learn what your level of exposure may be to certain chemicals in the environment, specifically chemicals called phthalates. Phthalate is the only chemical that will be measured.

Additional Information:

All information collected during this study will be kept strictly confidential, and will not contain any personal identifiable information such as your name, address, and/or telephone number. All the information will be will be given a code number. To protect confidentiality, DNA data will not be linked to participant identifiers. Only the researcher in charge of the study will have access to the code numbers and be able to link any information to you. All samples and DNA data will be destroyed within three years after the conclusion of the study.

Length of Study:

After the questionnaire is complete and the urine sample has been collected, your participation on this study will be over.

This is an investigational study. Up to 300 participants (150 from Baytown,TX and 150 from the rural lower Rio Grande Valley in Hidalgo County, TX) will take part in this study. All will be enrolled through M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women of Mexican American origin ages 18 to 40 years
2. Residing in Baytown or the lower Rio Grande Valley in Hidalgo County, Texas
3. Who have signed the informed consent
4. Individuals will have had to reside in the study area for at least 5 years
5. Pregnant women are eligible for the study.

Exclusion Criteria:

1) None

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men and Women of Mexican American origin ages 18 to 40 years, residing in Baytown or the lower Rio Grande Valley in Hidalgo County, Texas for at least 45 years.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-05-15 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of exposure to chemical/toxins (Survey Responses) | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Hajek, PHD, MS, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Goose Creek Consolidated Independent School District, Baytown, Texas
  - Texas Southern University, Houston, Texas
  - LaJoya Independent School District, La Joya, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org